CLINICAL TRIAL: NCT05038774
Title: Impact of Educational Intervention on Hypertension Management by Primary Care Physician (Pump)
Brief Title: Educational Intervention for Hypertension Management
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Karachi (Other)
Collaborators: Advanced Education & Research Center (Other)
Responsible Party: Principal Investigator, Prof. Dr. Tariq Ashraf, Principal Investigator, University of Karachi
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: PUMPKG
Record Dates: First submitted 2021-08-22; First posted 2021-09-09 (Actual); Last update posted 2021-09-17 (Actual); Status verified 2021-09

CONDITIONS: Hypertension
Keywords: Educational Intervention; Hypertension Management; Primary Care Physician
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventional group (Experimental): GPs of the Interventional group will receive (1 day) face to face education with structured educational material on strategies of hypertension management by a senior cardiologist.
  Interventions: Other: Face to face Educational Training
- Control group (Active Comparator): GPs of the Control group will receive print version of education material (Structured educational material) on strategies of structured hypertension management.
  Interventions: Other: Printed Education Material

INTERVENTIONS:
Other: Face to face Educational Training — 1. Key points of current hypertension guidelines.
  2. 10-step checklist how to obtain standardized upper arm blood pressure readings according to guidelines.
  3. template of a blood pressure documentation sheet for serial documentation of blood pressure values by patients.
  4. checklists to assist in the diagnosis of secondary hypertension.
  5. Patient information leaflet about hypertension.
  Arms: Interventional group
Other: Printed Education Material — 1. Key points of current hypertension guidelines.
  2. 10-step checklist how to obtain standardized upper arm blood pressure readings according to guidelines.
  3. template of a blood pressure documentation sheet for serial documentation of blood pressure values by patients.
  4. checklists to assist in the diagnosis of secondary hypertension.
  5. Patient information leaflet about hypertension.
  Arms: Control group

SUMMARY:
An interventional study is designed and a structured educational session will be conducted regarding the management of Blood pressure for the general physicians of Karachi, Lahore, Peshawar, Islamabad, Multan and Quetta. The purpose of designing this study is to observe the effect of hypertension educational intervention for general physicians to improve patient outcomes indirectly. Results of this study may provide a basis for developing a hypertension educational program targeted at general physicians.

DETAILED DESCRIPTION:
Study Procedure

1. Screening of General physicians as per inclusion criteria and recruitment of GPs by clinical research associate after obtaining informed consent form.
2. GPs will be asked to fill hypertension awareness questionnaire at baseline
3. Both group of GPs with the help of clinical research associate will recruit 5 patients from study site.
4. After obtaining informed consent, Patient will be asked to fill hypertension awareness questionnaire at baseline or recruitment day and share pictures of 12-hour blood pressure measurement (from digital BP apparatus) with clinical research associate.
5. Randomization of GPs will be than in to 2 Groups.
6. After randomization, Group 1 GPs will receive (1 day) face to face education and Group 2 GPs will receive print version of education material.
7. After GPs education intervention, patients will be invited for regular checkup at GPs clinic.
8. Patient will be again asked to fill hypertension awareness questionnaire after 3 months and share pictures of 12-hour blood pressure measurement (from digital BP apparatus) with clinical research associate. (1st, 2nd & 3rd Month).
9. GPs will be asked to fill hypertension awareness questionnaire again after 3 months (Post intervention)

ELIGIBILITY:
Inclusion Criteria:

* GPs who have at least three years of practice experience in the broad disciplines of primary care using the Numerical Pain Rating (NPR) scale over the past week ≥ 2 on a 0-10 numerical pain scale.
* Patients between 18-60 years.
* Patients with uncontrolled blood pressure according to Pakistan hypertension league guidelines
* Patients with or without angiographically proven coronary, peripheral or cerebral vascular disease.
* Patients must be able to give informed consent and be able to read and comprehend in the Urdu (National Language)
* Patients must have a digital BP apparatus at home.
* Patients must have a phone with camera and internet.

Exclusion Criteria:

* GPs who had attended a planned Hypertension educational program during the last 6 months.
* Patients with a recognized psychiatric disorder as per the Diagnostic and Statistical Manual of Mental Disorders

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 126 (Estimated)
Dates: Start 2021-09-30 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Blood Pressure | 3 Months
  Pre & Post change in the blood pressure control rate. Defined as percentage of patients with an average 12-hour blood pressure <130/80 mmHg.

SECONDARY OUTCOMES:
Knowledge of GPs about Hypertension Management | 3 Months
  Pre & Post knowledge enhancement of GPs regarding hypertension management.
Knowledge of Patients about Hypertension Management | 3 Months
  Pre & Post knowledge enhancement of patients regarding hypertension

CONTACTS AND LOCATIONS:
Locations (1):
- Karachi institute of heart disease, Karachi, Sindh, Pakistan

REFERENCES:
- [Background] Ezzati M, Lopez AD, Rodgers A, Vander Hoorn S, Murray CJ; Comparative Risk Assessment Collaborating Group. Selected major risk factors and global and regional burden of disease. Lancet. 2002 Nov 2;360(9343):1347-60. doi: 10.1016/S0140-6736(02)11403-6. PMID 12423980
- [Background] Lawes CM, Bennett DA, Feigin VL, Rodgers A. Blood pressure and stroke: an overview of published reviews. Stroke. 2004 Apr;35(4):1024. PMID 15053002
- [Background] Tu K, Chen Z, Lipscombe LL; Canadian Hypertension Education Program Outcomes Research Taskforce. Prevalence and incidence of hypertension from 1995 to 2005: a population-based study. CMAJ. 2008 May 20;178(11):1429-35. doi: 10.1503/cmaj.071283. PMID 18490638
- [Background] Marques-Vidal P, Tuomilehto J. Hypertension awareness, treatment and control in the community: is the 'rule of halves' still valid? J Hum Hypertens. 1997 Apr;11(4):213-20. doi: 10.1038/sj.jhh.1000426. PMID 9185025
- [Background] Primatesta P, Brookes M, Poulter NR. Improved hypertension management and control: results from the health survey for England 1998. Hypertension. 2001 Oct;38(4):827-32. PMID 11641294